CLINICAL TRIAL: NCT05084196
Title: Melatonin for the Prevention of Antibiotic Associated Acute Kidney Injury
Brief Title: Melatonin for Prevention of Kidney Injury
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Luigi Brunetti, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro2021001502
Record Dates: First submitted 2021-09-13; First posted 2021-10-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Acute Kidney Injury; Adverse Drug Event
MeSH Terms: conditions — Acute Kidney Injury; Drug-Related Side Effects and Adverse Reactions | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Melatonin Arm (Experimental): Melatonin 5 mg capsule by mouth at bedtime for the duration of hospitalization or discontinuation of broad spectrum antibiotics, whichever comes first.
  Interventions: Drug: Melatonin
- Placebo Arm (Placebo Comparator): Placebo capsule by mouth at bedtime for the duration of hospitalization or discontinuation of broad spectrum antibiotics, whichever comes first.
  Interventions: Other: Placebo Capsule

INTERVENTIONS:
Drug: Melatonin — Melatonin 5 mg capsule by mouth at bedtime
  Arms: Melatonin Arm
Other: Placebo Capsule — Placebo capsule by mouth at bedtime
  Arms: Placebo Arm

SUMMARY:
This study will evaluate the safety and effectiveness of melatonin for the prevention of antibiotic associated acute kidney injury in hospitalized patients.

DETAILED DESCRIPTION:
Consenting subjects meeting inclusion and exclusion will be randomized to receive melatonin 5 mg daily or a matching placebo. Study subjects will be followed for the duration of hospitalization or discontinuation of broad spectrum antibiotics (vancomycin plus piperacillin/tazobactam). The primary outcome and secondary outcomes will be evaluated by the study team.

ELIGIBILITY:
Inclusion criteria:

* Aged 18 to 75 years
* Currently prescribed vancomycin with the presumption that therapy will be continued for at least 3 days based on a review of subject status. Because of the critical nature of starting empiric broad-spectrum antibiotics, we will allow one dose of the antibiotic combination before consent and enrollment. This strategy is necessary for the ethical conduct of the study.

Exclusion criteria:

* Estimated creatinine clearance < 30 mL/min
* Liver impairment (liver enzymes > 3 times upper limit)
* Any history of allergy or contraindication to melatonin
* Pregnancy or breastfeeding
* Autoimmune disease
* Requiring vasopressors
* Requiring mechanical ventilation
* History of acute kidney injury in the past 30 days
* Inability to take oral medications
* Clinical evidence of significant unstable or uncontrolled illness which, in the opinion of the research team, could confound the results of the study or put the patient at undue risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury | From date of randomization until the date of first documented acute kidney injury or date of antibiotic discontinuation, whichever came first, assessed up to 28 days
  Acute kidney injury will be defined as an increase in sCr from baseline of >/= 0.3 mg/dL or a >/= 50% increase from baseline.

OTHER OUTCOMES:
Melatonin plasma trough concentration | Days 3, 5, and 7
  Evaluate the steady state plasma trough concentration of melatonin
Piperacillin/tazobactam plasma trough concentration | Days 3, 5, and 7
  Evaluate the steady state plasma trough concentration of piperacillin/tazobactam
Vancomycin plasma Area Under the Curve (AUC) | Days 3, 5, and 7
  Evaluate the steady state plasma AUC of vancomycin
Association between Kidney Injury Molecule-1 (KIM-1) and serum creatinine | Days 3, 5, and 7
  Measure KIM-1 in plasma and urine and evaluate discordance between serum creatinine.
Mitochondrial stress assessment via extracellular flux analysis to measure oxygen consumption rate of cells | Days 1 and 3
  Evaluate mitochondrial stress in peripheral blood mononuclear cells from a subset of subjects in each group. In addition, mitochondrial stress will be evaluated on day 3 in a subset in the melatonin group.
Urine mitochondrial DNA copy number | Days 1, 3, 5, and 7
  Measure mitochondrial DNA (mtDNA) in urine samples using polymerase chain reaction (PCR).
Fold-change in NRF-2 gene expression in peripheral blood mononuclear cells | Days 1 and 5
  Measure gene expression level at baseline and then on day 5 (or last day of study if earlier) using polymerase chain reaction (PCR) and compare the fold-change from baseline between groups.
Number of subjects with NRF2 DNA single nucleotide polymorphisms | Day 1
  Determination of the number of individuals with NRF2 DNA single nucleotide polymorphisms in the study population and compare the incidence of primary outcome in those with and without polymorphisms.
Number of subjects with KEAP1 DNA single nucleotide polymorphisms | Day 1
  Determination of the number of individuals with KEAP1 DNA single nucleotide polymorphisms in the study population and compare the incidence of primary outcome in those with and without polymorphisms.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Brunetti, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (2):
- United States (2):
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey

IPD SHARING:
Plan to Share IPD: No